CLINICAL TRIAL: NCT06683014
Title: The Effects of MDMA (3,4-methylenedioxymethamphetamine) in Social Cognition in Borderline Personality Disorder
Brief Title: MDMA in Borderline Personality Disorder
Acronym: MDMA in BPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Connecticut Mental Health Center (Unknown)
Responsible Party: Principal Investigator, Sarah Fineberg, Assistant Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000037769
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Borderline Personality Disorder
Keywords: 3,4-methylenedioxymethamphetamine; social cognition
MeSH Terms: conditions — Borderline Personality Disorder | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label MDMA (Experimental): Participants will receive one dose of open-label 3,4-methylenedioxymethamphetamine (MDMA).
  Interventions: Drug: MDMA

INTERVENTIONS:
Drug: MDMA — Participants will receive one dose of open-label 3,4-methylenedioxymethamphetamine (MDMA).
  Other Names: 3,4-methylenedioxymethamphetamine

SUMMARY:
The purpose of this study is to test the effects of MDMA (3,4-methylenedioxymethamphetamine) on social cognition in adults with Borderline Personality Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-60 years
* Body weight between 110 and 210 pounds. Minimum body mass index (BMI) 16.5.
* Able to swallow pills.
* Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable and must sign release of information for this contact person.
* People of childbearing potential must agree to utilize a highly effective method of birth control (including the following, in accordance with Clinical Trials Facilitation and Coordination Group (CTFG) guidelines: combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation, including oral, intravaginal, and transdermal administrations; estrogen-only hormonal contraception associated with inhibition of ovulation, including oral, injectable, and implantable forms; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; abstinence from sexual activity with biological males) and for one month prior to dosing and for the duration of the two week follow-up period.
* Able to provide written informed consent according to Yale IRB guidelines.
* Able to read and write English proficiently.
* Diagnosis of BPD, as determined by the Diagnostic Interview for Personality Disorders BPD questions (DIPD), including endorsement of the criteria for abandonment fears and for stormy relationships.
* No exposure to MDMA in the last 6 months, and no more than 10 lifetime uses of ecstasy.
* Agree not to drive a motor vehicle for 24 hours after the treatment day. Agree to identify a support person to accompany them home after the medication day.
* Are willing to remain overnight at the study site after each experimental session until the next morning if recommended by the study physician
* Currently not taking contraindicated medications (antidepressants, antipsychotics, mood stabilizers, stimulants).
* Medications not on the contraindicated list must be reviewed and approved by the study PI
* For people in mental health care, signs releases for the study investigators to communicate with their mental healthcare provider and medical doctor(s) about their medical and mental health history and their mental and medical status during the study. When contacted, the mental healthcare provider confirms the ongoing treatment relationship.
* For people not in mental health care acknowledges receipt of local resources for mental healthcare.
* For all participants, acknowledges receipt of local emergency resources

Exclusion Criteria:

* History of bipolar disorder, schizophrenia or schizoaffective disorder or currently exhibiting psychotic features as determined by the Structured Clinical Interview for DSM5 (SCID-5) and/or clinician assessment.
* Lifetime diagnosis of autism.
* Serious suicide risk in the past 6 months, as assessed by Columbia Suicide Severity Rating Scale (CSSRS) type 4 or 5 ideation, or suicidal behavior (CSSRS item) or preparatory acts (CSSRS item).
* Any current substance use disorder (in the last 1 month) per SCID interview for alcohol or non-alcohol substances; or a positive pre-study (screening) urine drug screen.
* Any severe substance use disorder during the last 6 months.
* Any significant history of serious medical or neurological illness (including history of stroke, myocardial infarction, heart failure, cardiac arrhythmia, diabetes, family history of long-QT syndrome, etc.)
* Any signs of major medical or neurological illness on examination, ECG screening, or laboratory tests. For QTc, we would exclude for QTcf >450. For liver function tests (AST, ALT), we will exclude for values more than 2.5 times the upper limit of normal range for our laboratory. For kidney function, we would exclude for eGFR < 90 (n.b. our laboratory does use the contemporary non-race based formula for eGFR). Clinically significant electrolyte imbalances (sodium, potassium values out of range) will also be exclusionary (clinical significance to be determined by study MD review). A participant with a clinical abnormality may be included only if the study physician considers the abnormality will not introduce additional risk factors and will not interfere with the study procedure.
* History of valvulopathy or pulmonary hypertension (due to evidence of 5HT2B receptor agonism by MDMA)
* History of uncontrolled hypertension with baseline blood pressure above 130 mmHg (systolic) and over 90 mmHg (diastolic). Any history of syncope and/or study baseline blood pressure below 90 mmHg (systolic).
* History of tachycardia with baseline heart rate above 90 beats per minute.
* Current pregnancy or breastfeeding as assessed by patient report or by urine pregnancy test.
* Taking any contraindicated medications: antidepressants, mood stabilizers, antipsychotics, stimulants. No patient will be encouraged to discontinue medications for the study. We will allow people to participate who stopped contraindicated medications at least five half-lives before baseline assessments.
* Hypersensitivity to non-MDMA ingredients of the investigational medicine product (IMP), namely mannitol, magnesium stearate, and hydroxypropylmethylcellulose.
* Herbal and dietary supplements will be reviewed on a case-by-case basis by the sponsor-PI for decision about safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Reported Social Cognition After 1 Dose of MDMA. | From baseline (immediately before drug dose) to 2 hours after drug dose on the same day.
  Defined as sociability visual-analogue scale (VAS) score. Total score range is 0-100, higher scores indicating more sociability.

SECONDARY OUTCOMES:
Change from baseline in emotion appraisal on facial emotion recognition task score, on same day after drug administration. | From baseline (immediately before drug dose) to 2 hours after drug dose on the same day.
  The facial-emotion recognition task is a computer-based cognitive task for measuring ability to recognize facial emotions, that yields accuracy scores for positive and negative emotions. Possible scores range from 0 (poor facial emotion recognition) to 100% (excellent facial emotion recognition).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Fineberg, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share to share individual participant data.